CLINICAL TRIAL: NCT05534555
Title: Point of Care Testing Using FebriDx to Improve Antibiotic Use for Respiratory Tract Infections in Primary Care: a Mixed Methods Feasibility Study
Brief Title: Point of Care Testing Using FebriDx in Primary Care: a Mixed Methods Feasibility Study
Acronym: PREFIX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 72411
Record Dates: First submitted 2022-06-08; First posted 2022-09-09 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Lower Resp Tract Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Febridx (Other): Undergo FebriDx testing
  Interventions: Diagnostic Test: FebriDx

INTERVENTIONS:
Diagnostic Test: FebriDx — Testing of finger-prick blood sample using FebriDx

SUMMARY:
This is a mixed-methods, multi-centre feasibility study. Formal advice and peer-review with regards to study design was sought from the Southampton Research Design Service (RDS), the NIHR CRN Wessex, and patient contributors during the development of the grant application. We will recruit up to ten GP practices, each given 20-40 FebriDx tests (300 in total). Up to four clinicians per practice will be trained to use the test. A sequential explanatory approach to data collection will be taken (21), with quantitative data analysis in stage one, followed by qualitative interviews with the study's practice participants in stage two.

DETAILED DESCRIPTION:
It can be difficult to tell the difference between viral and bacterial infections. Many patients are therefore prescribed antibiotics unnecessarily. Overuse of antibiotics is leading to a crisis of 'antibiotic resistance', where antibiotics no longer work for some infections.

FebriDx ® is a new hand-held test that uses a 'finger-prick' of blood, and within 10 minutes, provides a result that can help clinicians decide whether an infection is likely to be caused by a virus or bacteria. This could help clinicians decide when antibiotics are needed, but the test has not been adequately tested in primary care.

We would like to do a future study to test whether FebriDx can safely reduce antibiotic prescriptions in primary care.

However, before we do this, we need to do a smaller 'feasibility' study to explore how easy to use the FebriDx test is and, what GPs and patients think of the test, and to help us design a larger future study.

Aims

1. Explore whether FebriDx could reduce the use of antibiotics for chest infections in primary care.
2. Explore how feasible it would be to do a large research study in the future using FebriDx

Methods

We will recruit up to ten GP practices, each given 20-40 FebriDx tests (300 total).

Stage one Patients with a chest infection will be invited to participate if their clinician has decided that they are likely to prescribe antibiotics. Following consent, the clinician will record some basic information about the patient, and the patient will undergo the FebriDx test. The clinician will then record whether or not they prescribed antibiotics and if they think the test had an effect on their decision. Patients will also undergo an optional nasopharyngeal swab.

Stage two Clinicians and patients will be interviewed on how useful they think FebriDx testing is, and how they think we should design a larger future study.

ELIGIBILITY:
Inclusion Criteria:

* Lower respiratory tract infection (defined as in previous studies as an acute cough as the predominant symptom, judged by the GP to be infective in origin, lasting <21 days, and with other symptoms or signs localising to the lower respiratory tract (shortness of breath, sputum, chest pain). This is a definition which we have used in previous studies (22)
* The clinician has decided that they are likely to prescribe antibiotics in the absence of further diagnostic testing
* The patient is at the surgery or willing to attend the surgery for a face-to-face assessment
* The patient (or their parent or legal guardian) can follow the study procedures and is willing to provide informed consent

Exclusion Criteria:

* Patients who have taken antibiotics within the last 30 days
* Participant (or their parent/guardian) unable to provide informed consent

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Six months
  The proportion of patients recruited as compared to the number invited to participate
Antibiotic prescription rate at study visit | At study visit (baseline)
  The proportion of patients prescribed antibiotics at the study visit
Antibiotic prescription rate over entire study period | Within 30 days of recruitment
  The proportion of patients prescribed antibiotics within 30 days of recruitment
Test failure rate | After FebriDx use (baseline)
  The proportion of Febridx tests which fail to provide a valid result
Ease-of-use scores | Six months
  The average ease-of-use score for the device as determined by users.
  Each user will be asked to grade the device according to a modified US Clinical Laboratory Improvement Amendments (CLIA) categorisation criteria
  Within each of the 11 categories, a score of '1' indicates the lowest level of complexity, and the score of '3' indicates the highest level, to derive a measure of complexity (total score range 1 - 33)
Subsequent healthcare contacts | Within 30 days of recruitment
  The proportion of patients undergoing subsequent healthcare contact
Subsequent serious complication rate | Within 30 days of recruitment
  The proportion of patients undergoing significant complications (sepsis, ITU admission, or death)

SECONDARY OUTCOMES:
FebriDx sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) for diagnosis of viral infection | Within one year
  FebriDx sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) for diagnosis of viral infection, as determined by comparison of FebriDx result with nasopharyngeal swab analysis by gold-standard viral PCR

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Wilcox, Principal Investigator — University of Southampton

IPD SHARING:
Plan to Share IPD: No